CLINICAL TRIAL: NCT01947829
Title: Interdialytic Kt/V Variability Measurement With Adimea (IVP STUDY)
Acronym: IVP
Status: Completed | Type: Observational
Sponsor: B.Braun Avitum AG (Industry)
Responsible Party: Sponsor
Other Study IDs: BA-O-H-1205
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Kidney Disease
Keywords: hemodialysis; dialysis dose
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Hemodialysis

SUMMARY:
Session-to-session variations in delivered Kt/V that may cause failure to achieve the prescribed dialysis dose may be significant in regular clinical practice. To date, this is not recognized due to monthly blood Kt/V measurements only. Suboptimal delivery of prescribed dialysis dose may be caused by low effective treatment time, vascular access dysfunction, hemodynamic stability, blood pump speed, membrane influences, lab value variability or others which may vary from session to session. Patients close to recommended target limits of dialysis dose may thus be "randomly" attributed to be adequately or inadequately dialyzed. Therefore, in the literature, use of average Kt/V values is recommended.

Adimea allows easy Kt/V determination in every session and thus documentation of the monthly achieved Kt/V in patients who repeatedly miss Kt/V. Knowledge, therefore, of session-to-session variability as well as knowledge of dialysis dose monitoring at every dialysis may enhance and secure delivery of adequate dialysis.

The main objective is the estimation of the pooled within-patient SDs (standard deviation) for single treatment Adimea and of urea kinetic modeling (UKM)/ blood spKt/V. Failure of Kt/V>1.2 delivery as well as its potential causes will be assessed. spKt/V target achievement is assessed by monitoring dose by Adimea at every dialysis. This shall demonstrate that session-to-session variability can be decreased with usage of Adimea.

ELIGIBILITY:
Inclusion Criteria:

* Patient on chronic hemodialysis for at least 6 months
* Thrice dialysis therapy weekly
* Stable fistula access
* Documented three, monthly blood spKt/V from 1.0 to 1.4 or
* Average of spKt/V<1.35 out of three consecutive blood measurements
* Age ≥ 18 years
* Voluntary participation and written informed consent

Exclusion Criteria:

* Severe hematologic disorders (e.g. multiple myeloma)
* Life expectancy less than 6 months
* Single-needle dialysis
* Patient was monitored with Adimea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on chronic hemodialysis.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Dialysis dose (spKt/V) measured by Adimea and Urea Kinetic Modeling (UKM) | Six months prospective

SECONDARY OUTCOMES:
Treatment time | Six months prospective
  Dialysis time per session
Blood flow rate | 6 months prospective
  Initial blood flow rate [ml/min] at the beginning of dialysis session.
Dialysate flow rate | 6 months prospective
  Initial dialysate flow rate [ml/min] at the beginning of dialysis session.
Ultrafiltration volume | 6 months prospective
  Ultrafiltration volume [ml] reached at the end of dialysis session.
Dialyser size | 6 months prospective
  Membrane surface size [m2] of the dialyser used during dialysis session.
Hemoglobin | 6 months prospective
  Hemoglobin level [mmol/l or g/dl] before dialysis.
Hematocrit | 6 months prospective
  Hematocrit level [%] before dialysis.
Intact parathyroid hormone (iPTH) | 6 months prospective
  Intact parathyroid hormone level [pmol/l or ng/l] before dialysis.
C-reactive protein (CRP) | 6 months prospective
  C-reactive protein level [mg/l or g/dl] before dialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangmei Chen, Prof., Principal Investigator — China PLA General Hospital (301 hospital)
Locations (2):
- China (2):
  - Beijing Friendship Hospital,Capital Medical University, Beijing
  - China PLA General Hospital (301 hospital), Beijing